CLINICAL TRIAL: NCT01930708
Title: A Multicenter, Open-Label Study Evaluating the Effectiveness of Oral Tecfidera™ (Dimethyl Fumarate) on MS Disease Activity and Patient-Reported Outcomes in Subjects With Relapsing-Remitting Multiple Sclerosis in the Real-World Setting
Brief Title: A Study Evaluating the Effectiveness of Tecfidera (Dimethyl Fumarate) on Multiple Sclerosis (MS) Disease Activity and Patient-Reported Outcomes
Acronym: PROTEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109MS408; 2013-001656-35 (EudraCT Number)
Record Dates: First submitted 2013-08-15; First posted 2013-08-29 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis
Keywords: BG-12
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DMF (Experimental): 120 mg capsule oral twice daily (BID) during the first week and 240 mg BID thereafter.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — Administered as per the approved dosage in all countries where DMF has received marketing authorization.
  Other Names: Tecfidera; DMF; BG00012

SUMMARY:
The primary objective of the study is to estimate the annualized relapse rate (ARR) in participants with Relapsing Remitting Multiple Sclerosis (RRMS) who are treated with dimethyl fumarate (DMF) over a 12-month period.

The secondary objectives of this study in this population are to assess the impact of DMF over a 12-month period on participants -reported health-related quality of life (HRQoL) outcomes, additional clinical effectiveness outcomes, and health economics-related outcomes, and to characterize participants-reported adherence to DMF.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a diagnosis of Relapsing-Remitting Multiple Sclerosis (RRMS) and satisfy the approved therapeutic indication for DMF (per the local DMF product information).
* Must be naïve to DMF, Fumaderm®, and other compounded fumarates, and to MS therapies that are primarily prescribed second-line (e.g., natalizumab, fingolimod) and to alemtuzumab.
* Have a recent complete blood count (CBC) that does not preclude the subject's participation in the study, in the judgment of the Investigator.

Key Exclusion Criteria:

* Are unwilling or unable to comply with study requirements, or are deemed unsuitable for study participation as determined by the Investigator.
* Have major comorbid conditions that preclude participation in the study, as determined by the Investigator.
* Are pregnant, unless DMF is clearly needed and the potential benefit of DMF to the subjects justifies the potential risk to the fetus, in the judgment of the Investigator (in all countries except Austria). In Austria, pregnant subjects are excluded from participation in the study.
* Are women of childbearing potential and are not using appropriate contraception (per the local DMF product information) as determined by the Investigator.
* Women who are breastfeeding may be excluded (per the local DMF product information) at the discretion of the Investigator.
* Have previously received or are receiving treatment with MS therapies primarily used second-line (e.g., natalizumab, fingolimod) or alemtuzumab, or are currently receiving and planning to continue on other disease-modifying therapies for RRMS.
* Are hypersensitive to the active ingredient in the DMF drug product (i.e., DMF) or to any of the excipients listed in the local DMF product information.
* Current enrollment in any clinical trial except for the Biogen Idec DMF Pregnancy Exposure Registry or other studies that, according to the study Medical Director, do not conflict with this study (e.g., health economics studies or local registries).

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1114 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | 12 Months

SECONDARY OUTCOMES:
Change from Baseline in Multiple Sclerosis Impact Scale (MSIS-29) score | 12 Months
  This is a validated, 29-item, MS-specific HRQoL scale that measures the physical (20 items) and psychological (9 items) impact of MS on the participant's day-to-day life during the previous 2 weeks. For each item, the subject is asked to circle the number that best describes his or her situation. The numbers for each item range from 1 (not at all) to 5 (extremely).
Change from Baseline in Modified Fatigue Impact Scale-5 Item (MFIS-5) score | 12 Months
  This scale consists of 5 statements that describe how fatigue may affect a person. For each statement, the participant is asked to circle the number that best indicates how often fatigue has affected him or her during the previous 4 weeks. The numbers for each question range from 0 (never) to 4 (almost always).
Change from Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) score | 12 Months
  This is a validated, 14-item questionnaire that measures a participant's level of satisfaction/dissatisfaction with medication.
Change from Baseline in EQ-5D 5 level version (EQ-5D-5L) index | 12 Months
  The widely validated EQ-5D includes 2 components, the EQ-5D descriptive system and the EQ VAS. The EQ-5D descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the subject is instructed to indicate whether he or she has "no problems" (level 1), "slight problems" (level 2), "moderate problems" (level 3), "severe problems (level 4), or "extreme problems/inability" (level 5) on that day. For the EQ VAS, the participant is instructed to mark an "x" on a vertical scale at the point that best describes his or her own health on that day, where 0 represents the "worst health" he or she can imagine and 100 the "best health" he or she can imagine.
Change from Baseline in participants-Reported Indices for Multiple Sclerosis-Activity Limitations (PRIMUS-Activity Limitations) score | 12 Months
  This 15-item component of the PRIMUS assesses a participant's ability to carry out various activities of daily living during the previous week without the use of aids (e.g., cane, walker, or wheelchair) or assistance. For each item, the participant is asked whether he or she can perform the activity without difficulty or with difficulty, or is unable to perform the activity.
Change from Baseline in Work Productivity and Activity Impairment-Multiple Sclerosis version (WPAI-MS) score | 12 Months
  This 6-item instrument assesses employment status, and, during the previous 7 days, hours of missed work due to MS or other reasons, hours worked (if employed), effect on productivity due to MS while working, and activity impairment attributable to health problems.
Change from Baseline in Beck Depression Inventory-Fast Screen (BDI-Fast Screen) score | 12 Months
  This is a 7-item scale that evaluates depression in participants with medical illness during the prior 2 weeks. It has been validated in subjects with MS.
Proportion of participants with confirmed (24-week) Expanded Disability Status Scale (EDSS) progression | 12 Months
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Annualized Relapse Rate (ARR) at Baseline (i.e., over the 12 months prior to enrollment) and at Month 6 | Baseline, 6 Months
The proportion of participants relapsed | 12 Months
Number of participants who are hospitalized/have emergency room visits due to MS relapses or have relapses requiring intravenous (IV) steroid treatment during the study, or who make visits to neurologists/other specialists due to MS | 12 Months
Proportion of participants who are hospitalized/have emergency room visits due to MS relapses or have relapses requiring intravenous (IV) steroid treatment during the study, or who make visits to neurologists/other specialists due to MS | 12 Months
Proportion of participants who report taking the prescribed DMF dose | 12 Months
Percentage of participants who report taking the prescribed DMF dose | 12 Months
Reasons reported by participants for not taking prescribed DMF dose | 12 Months
Change from baseline in EQ Visual Analog Scale (EQVAS) score | 12 Months
  A component of the EQ-5D, where participants are asked to rate their overall health-related quality of life on a standard vertical 20 cm visual analogue scale (similar to a thermometer) between 100 (best health imaginable) and 0 (worst health imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (83):
- Austria (7):
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Vienna
  - Research Site, Villach
- Belgium (3):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Melsbroek
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, Saint John's, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
- Czechia (6):
  - Research Site, Brno
  - Research Site, Havířov
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Pardubice
  - Research Site, Prague
- France (18):
  - Research Site, Strasbourg, Bas Rhin
  - Research Site, Dijon, Cote dÝOr
  - Research Site, Besançon, Doubs
  - Research Site, Nîmes, Gard
  - Research Site, Bordeaux, Gironde
  - Research Site, Colmar, Haut Rhin
  - Research Site, Toulouse, Haute Garonne
  - Research Site, Limoges, Haute Vienne
  - Research Site, Rennes, Ille Et Vilaine
  - Research Site, Grenoble, Isere
  - Research Site, Nantes, Loire Atlantique
  - Research Site, Reims, Marne
  - Research Site, Lille, Nord
  - Research Site, La Roche-sur-Yon, Vendee
  - Research Site, Poitiers, Vienne
  - Research Site, Le Chesnay, Yvelines
  - Research Site, Nancy
  - Research Site, Rouen
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Veszprém
- Italy (14):
  - Research Site, Ancona
  - Research Site, Bergamo
  - Research Site, Bolzano
  - Research Site, Castelfiorentino
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Perugia
  - Research Site, Pozzilli
  - Research Site, Roma
  - Research Site, Siena
  - Research Site, Torino
- Portugal (7):
  - Research Site, Almada
  - Research Site, Amadora
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Porto
  - Research Site, Setúbal
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Prešov
- Slovenia (2):
  - Research Site, Ljubljana
  - Research Site, Maribor
- Spain (11):
  - Research Site, Majadahonda, Madrid
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Córdoba
  - Research Site, El Palmar
  - Research Site, Girona
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vigo
  - Research Site, Zaragoza

REFERENCES:
- [Derived] Berger T, Brochet B, Brambilla L, Giacomini PS, Montalban X, Vasco Salgado A, Su R, Bretagne A. Effectiveness of delayed-release dimethyl fumarate on patient-reported outcomes and clinical measures in patients with relapsing-remitting multiple sclerosis in a real-world clinical setting: PROTEC. Mult Scler J Exp Transl Clin. 2019 Dec 2;5(4):2055217319887191. doi: 10.1177/2055217319887191. eCollection 2019 Oct-Dec. PMID 31832225